CLINICAL TRIAL: NCT00901550
Title: The Chinese University of Hong Kong Early Arthritis Study
Acronym: ERA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai-Shan Tam, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERA_2008
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Rheumatoid Arthritis
Keywords: MTX; anti-TNF; Early RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methotrexate (Active Comparator): A drug for RA patient
  Interventions: Drug: Methotrexate
- Infliximab (Active Comparator): for RA treatment
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Methotrexate — All participants received oral Methotrexate(MTX), starting at 7.5 mg/week. In patients with persistent tender or swollen joints, the dose was escalated in a graduated manner (2.5 mg/week every 1-2 weeks) to 15 mg/week by week 4 or 20 mg/week by week 8
  Other Names: MTX
  Arms: Methotrexate
Drug: Infliximab — Patients in combination group receive infliximab 3mg/kg at weeks 0, 2, and 6 and every 8 week thereafter.
  Other Names: Remicade
  Arms: Infliximab

SUMMARY:
The purpose of this study is:

1. To ascertain whether the quantitative assessment of enhancing synovial volume and perfusion indices on serial Magnetic Resonance Imaging (MRI) examination are useful indicators of responsiveness to treatment in early Rheumatoid Arthritis (RA) using biologic therapy and Methotrexate (MTX) compared with Methotrexate(MTX) alone.
2. To assess the cost-effectiveness of Tumor Necrosis Factor (TNF) blockers compared with Methotrexate(MTX) monotherapy for Rheumatoid Arthritis(RA).

DETAILED DESCRIPTION:
This was a 24-week open-label randomized study. Forty patients are randomly assigned to receive either combination infliximab plus Methotrexate(MTX) (n=20) or Methotrexate(MTX) alone (n=20)

All participants received oral Methotrexate(MTX), starting at 7.5 mg/week. In patients with persistent tender or swollen joints, the dose was escalated in a graduated manner (2.5 mg/week every 1-2 weeks) to 15 mg/week by week 4 or 20 mg/week by week 8 Patients in combination group receive infliximab 3mg/kg at weeks 0, 2, and 6 and every 8 week thereafter. Comprehensive assessment will be made on week 0, 12, 24.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 years of age or older
* Clinical diagnosis of RA with a duration not more than 24 months (Fulfilled the 1987 American College of Rheumatology (ACR) criteria for RA)
* Patients at risk of developing persistent or erosive arthritis
* DAS 28 ≥ 3.2
* Prednisolone < 10mg/day and started at least 4 weeks before baseline
* Either has ESR ≥ 28, CRP ≥ 10, presence of rheumatoid factor or anti-CCP, present of HLADRB*0401 or DRB1*0404, and radiographic erosions
* Informed consent

Exclusion Criteria:

* Little or no ability for self-care
* Previous treatment with DMARDs other than antimalarials
* Concomitant treatment with an experimental drug
* Malignancy within the last 5 years
* Bone marrow hypoplasia
* Clinically significant renal disease ( serum creatinine level ≥ 150µmol/L) or estimated creatinine clearance > 75ml/min, alanine aminotransferase (ALT) exceeds the upper limit of normal
* History of any clinically significant adverse reaction to murine or chimeric proteins
* History of TB in the last 5 years
* Known to have hepatitis B, or hepatitis C
* Had an opportunistic infection (e.g. herpes zoster, cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 6 months before screening
* History or ongoing chronic or recurrent disease; renal infection, chest infection, urinary tract infection, ulcer or skin wound
* History of infected joint prosthesis and use of antibiotics for the joint
* Received intravenous antibiotics within 30 days or oral antibiotics within 14 days for screening
* History of known demyelinating diseases (multiple sclerosis or optic neuritis)
* Current signs or symptoms of severe diseases (renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurologic, etc)
* History or concurrent CHF
* History of lymphoproliferative disease, splenomegaly
* Female of childbearing potential, unwilling to use adequate contraception during the study
* Current or recent ( within the past 3 months) pregnancy and cancer
* Active smoker, alcohol or drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Changes in the volume of enhancing synovitis measured by Magnetic Resonance Imaging(MRI) as it corresponds to active, inflamed tissue and is therefore expected to be a better marker of disease activity. | week 24

SECONDARY OUTCOMES:
changes in the synovitis grading and the perfusion indices | 24 week
proportion of patients achieving ACR and EULAR responses | week 24
Correlation between the Magnetic Resonance Imaging(MRI) findings and changes on x-ray | week 24

CONTACTS AND LOCATIONS:
Overall Officials: Edmund K Li, MD, Principal Investigator — Chinese University of Hong Kong
Locations (3):
- China (3):
  - Department of Medicine and Therapeutics, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - The Prince of Wales Hospital, Hong Kong